## 1.2 SUNRISE TRIAL CONSENT FORM

<u>Title of research:</u> Scaling Up Nurturing care, a Radio Intervention to Stimulate Early child development in Burkina Faso: SUNRISE Cluster Randomised Control Trial (CRT)

## **Investigators**

Prof Betty Kirkwood. London School of Hygiene & Tropical Medicine (LSHTM), <u>betty.kirkwood@lshtm.ac.uk</u> (Chief Investigator)

Dr Zelee Hill, University College London (UCL), z.hill@ucl.ac.uk

Professor Pasco Fearon, UCL, p.fearon@ucl.ac.uk

Dr Jolene Skordis-Worrall, UCL, j.skordis @ucl.ac.uk

Mr Roy Head, Development Media International (DMI), roy@developmentmedia.net

Mr Bassirou Kagone, Head of DMI Burkina Faso Office, Bassirou.Kagone@developmentmedia.net

## **For more information contact:**

Sabin Lazare Dandjinou, +226 70 65 55 40 or sabindandjinou@yahoo.fr (SUNRISE field coordinator), or

Achille Mignondo Tchibozo, + 226 25 37 68 98 (office) or atchibozo@poverty-action.org (Research manager, IPA Francophone West Africa)

Thank you for considering taking part in this research. Please let me know if you consent to each element of the research that I will now read out:

## Please circle 'yes' or 'no' for all statements:

| Consent statements | Response | |
|---|---|---|
| I confirm that I have read the information sheet and/or have been given a clear explanation of the study and have had the opportunity to ask questions which have been answered to my satisfaction. | Yes | No |
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving a reason, and if I decide to withdraw, any personal information I have provided up to that point will be deleted unless I agree otherwise. | Yes | No |
| I understand that all personal information will be kept confidential by the project staff and that all efforts will be made to ensure I cannot be identified. | | No |
| I understand that I will not benefit directly from this study or from any possible outcome it may result in in the future. | Yes | No |
| I agree to respond to questions about myself, my family and my baby in today's interview. | | No |
| I understand that I will receive 11 further visits from you every three months when you will ask me more detailed questions about what my baby is able to do. | | No |
| I also understand that you will request permission to observe my child doing different things at the visit when they are 18-20 months old and at the final visit when they will be 30-32 months of age, and that you will give me more detailed information about these at the time of these visits and request my consent. | | No |
| I am happy for my responses to be recorded on a tablet or paper. | Yes | No |
| I am happy for you to write about what I say during the interviews in reports, on the understanding that you will not reveal my identity. | Yes | No |

| Consent statements | Response | |
|---|---|---|
| I am happy for you to include quotations from the interviews in reports, on the understanding that I will not be able to be identified from these quotes. | Yes | No |
| I am happy for the information collected during the visits to be transferred to London, UK. | Yes | No |
| I am happy for the information I provide to be used by others for future research. I understand that this will not include my name or any way of identifying me. | Yes | No |

| Name: | Husband/partner's name: |
|---|---|
| Village name: | Cluster name: |
| Household number: | Serial number: |
| <del></del> | <u></u> |
| Date | Signature or thumb print (circle which one) |
| *IF THE MOTHER IS LESS THAN 18 YEARS OF AGE (Countersigned by Husband/Parent): | |
| Husband / parent: Date, Printed name & signature or thumbprint (circle which one) | |
| **IF THE MOTHER IS UNABLE TO READ OR WRITE (Countersigned by Impartial Witness): | |
| Impartial witness: Date, Printed name | e & signature |
| <u>Interviewer statement</u> : I, the undersigned, attest that I have explained to the participant in a language she/he understands, the procedures to be followed in the research study and the risks and benefits involved, and that | |
| she has freely given her consent to participate (** in the presence of the above named impartial witness, where applicable). | |
| Date | Name & Signature of interviewer |